CLINICAL TRIAL: NCT06052553
Title: The Effectiveness of a Novel Neck Training Device on Objective Neck Strength and Cognitive Measures in Junior A Hockey Players
Brief Title: A Study of TopSpin360 Training Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mario Hevesi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-005197
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Ice Hockey

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (No Intervention): Subjects will receive no intervention for the duration of the hockey season.
- TopSpin360 Intervention Group (Experimental): Subjects will use TopSpin360, twice- weekly and use for the duration of the hockey season.
  Interventions: Device: TopSpin360

INTERVENTIONS:
Device: TopSpin360 — Helmet training device used to train head to stay stable during jarring impacts through dynamic and multi-planar neck strengthening.
  Arms: TopSpin360 Intervention Group

SUMMARY:
This research is being done to investigate the novel neck strengthening device, TopSpin360 and its effectiveness on measures of neck strength and cognitive function.

DETAILED DESCRIPTION:
The neck plays a very important role in head positioning, stabilization, and decrease risk and severity. Neck extension strength measure has been associated with a decrease in concussion risk in male rugby players. Neck muscle characteristics may play a vital role in mitigating head accelerations due to contact thus reducing head impact severity. We hypothesize enhanced neuromuscular characteristics of cervical muscles will decrease brain impairments due to repeated contact.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English Speaker.
* Medically cleared to play ice hockey.

Exclusion Criteria:

* Clinically documented hearing issues.
* In-ear hearing aid or cochlear implant.
* Implanted pacemaker or defibrillator.
* Metal or plastic implants in skull. lack of verbal fluency in the English language.
* History of seizures.
* Allergy to rubbing alcohol or EEG gel.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in peak force | Baseline, post-season (approximately 6 months)
  Measured by a neck isometric device, maximal load in kilograms that could be applied to head before deviation from neutral position.
Change in normalized peak force | Baseline, post-season (approximately 6 months)
  Measured by a neck isometric device, peak force divided by participant weight in kilograms.
Change in force steadiness | Baseline, post-season (approximately 6 months)
  Measured by a neck isometric device, average peak force.
Change in rate of force development (RFD) | Baseline, post-season (approximately 6 months)
  Automatically collected by the TopSpin360 device, the multi-planar rate of force development (RFD) in pounds of force per second collected in both clockwise and counterclockwise.
Change in visuo-motor reaction time | Baseline, post-season (approximately 6 months)
  Measured by a neck isometric device, reported in milliseconds (ms)
Change in blood biomarker levels | Baseline, post-season (approximately 6 months)
  Blood will be at a biomarker level. We will investigate 5 different markers: NfL, SNCB, vWF, SNCA, and BDNF. Each biomarker will be measured in Nanograms per Milliliter (ng/ml).
Change in salivary biomarkers | Baseline, post-season (approximately 6 months)
  Salivary biomarkers are relatively new and we will investigate to see if NfL, SNCB, vWF, SNCA, and BDNF. Each biomarker will be measured in Nanometer per milliliter (ng/ml).
Change in N100 Amplitude | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity N100 potential amplitude. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores.
Change in N100 Latency | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity N100 potential latency. Increased latencies are indicative of slower responses. Obtained by EEG recording of N100 potential amplitude. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores.
Change in P300 Amplitude | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity P300 potential amplitude. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores.
Change in P300 Latency | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity P300 potential latency. Increased latencies are indicative of slower responses. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores
Change in N400 Amplitude | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity N400 potential amplitude. Increased amplitudes are indicative of larger signals. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores.
Change in N400 Latency | Baseline, post-season (approximately 6 months)
  Electroencephalograph (EEG) recording of brain electrical activity N400 potential latency. Increased latencies are indicative of slower responses. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores.

SECONDARY OUTCOMES:
Change in King-Devick Test (KDT) scores | Baseline, post-season (approximately 6 months)
  A rapid number-naming test that requires individuals to read 3 numbered patters aloud as fast as possible, the resulting time if the KDT score. The post-season score is compared to the pre-season baseline. An increase in the number of seconds required to read the 3 number patterns is considered to be significant.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Hevesi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No